CLINICAL TRIAL: NCT05665621
Title: The Effect of Strength and Combined Balance Training Intervention Programme on Physical Function, Physical Activity, and Musculoskeletal Health in Children With Overweight and Obesity
Brief Title: The Effects of Strength and Balance Training on Physical Function in Overweight Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Mary's University, Twickenham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: StMarysUC7
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): Eight-week in-school strength and balance training program
  Interventions: Other: Eight-week in-school strength and balance training program
- Control (No Intervention): No intervention, normal activities.

INTERVENTIONS:
Other: Eight-week in-school strength and balance training program — Training program consisting of two 1-hour strength and balance training sessions per week.
  Arms: Training group

SUMMARY:
This intervention study aims to examine the efficacy of a school-based exercise programme to improve strength and balance in overweight and obese 7-11-year-olds in the United Kingdom. The main question[s] it aims to answer are:

* Is the school-based exercise programme effective in improving lower limb muscular strength and balance control?
* How do increases in strength and balance skills impact physical function, the risk to musculoskeletal health, and physical activity? Participants will attend baseline, post-intervention, and follow-up testing that includes assessment of strength, balance, 3D gait, plantar pressure, physical function and physical activity. The intervention group will take part in physical activity sessions in their school for 1 hour twice a week for a total of 8 weeks.

Researchers will compare the intervention group to a control group that will take part in no-activity sessions and carry out their normal school and seasonal activities.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese

Exclusion Criteria:

-

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-03-13 (Estimated); Primary Completion 2023-08-13 (Estimated); Study Completion 2023-08-13 (Estimated)

PRIMARY OUTCOMES:
Change in Body Mass Index Z-Score | Baseline to end of the 8-week intervention and to end of 8-week follow-up period.
  Body mass index will be calculated as body mass (kg) / height (m)2. Body mass will be measured using weighing scales and height by stadiometer whilst participants are barefooted with simple clothing (shorts and t-shirt). Z-scores denote the standard deviations that BMI for gender and height are from the mean of United Kingdom child reference curves. A higher z-score means greater BMI than the mean for child gender and height.
Change in body fat percentage | Baseline to end of the 8-week intervention and to end of 8-week follow-up period.
  Bioelectrical impedance will be used to determine whole-body impedance. Population-specific equations will be applied to estimate body fat (kg). The percentage of body fat will be calculated as (Fat Mass (kg)/Body Mass(kg))*100.
Change in fat free mass (kg) | Baseline to end of the 8-week intervention and to end of 8-week follow-up period.
  Bioelectrical impedance will be used to determine whole-body impedance. Population-specific equations will be applied to estimate body fat (kg). Fat-free mass will be calculated as Body Mass (kg) - fat mass (kg).
Change in lower limb 3D gait. | Baseline to end of the 8-week intervention and to end of 8-week follow-up period.
  Joint angles, moments, and power waveforms of hip, knee and ankle in three dimensions during the stance phase of self-paced walking. Change in lower limb 3D gait will be determined via a previously validated marker set for obese children, time normalised to 100% of stance phase, and moment and power will be dimensionless normalised to body mass and leg length.
Change in 3D foot in gait. | Baseline to end of the 8-week intervention and to end of 8-week follow-up period.
  The angle of the forefoot, midfoot, rearfoot and shank in three dimensions during the stance phase of self-paced walking. Change in foot 3D gait will be determined via a previously validated marker set for obese children, and time normalised to 100% of the stance phase.
Change in lower limb muscular strength relative to body mass. | Baseline to end of the 8-week intervention and to end of 8-week follow-up period.
  Isokinetic dynamometry will be used to determine the maximal strength of hip extension, hip flexion, hip adduction, hip abduction, knee extension, knee flexion, ankle plantarflexion, and ankle dorsiflexion. Maximal moments will be allometrically scaled to body mass.
Change in lower limb muscular strength relative to fat free mass. | Baseline to end of the 8-week intervention and to end of 8-week follow-up period.
  Isokinetic dynamometry will be used to determine the maximal strength of hip extension, hip flexion, hip adduction, hip abduction, knee extension, knee flexion, ankle plantarflexion, and ankle dorsiflexion. Maximal moments will be allometrically scaled to fat-free mass.
Change in six minute walk distance. | Baseline to end of the 8-week intervention and to end of 8-week follow-up period.
  The maximal distance walked in six minutes will be recorded in meters.
Change in sit to stand repetitions | Baseline to end of 8-week intervention and to end of 8-week follow up period.
  The maximal number of times participants are able to stand up and sit down in one minute. The stool used will be adjusted so the participant's knee is at 90 degrees when seated, and arms will be placed across the chest.
Change in timed up and go time | Baseline to end of the 8-week intervention and to end of 8-week follow-up period.
  The time (seconds) it takes participants to stand from seated (knees 90 degrees), arms across chest, walk 3m turn and go back to seating.
Change in single leg stance time | Baseline to end of the 8-week intervention and to end of 8-week follow-up period.
  The maximum amount of time participants are able to maintain stance on their dominant limb with the non-dominant limb flexed 90 degrees and hands held on the waist. The test is stopped when the non-dominant limb touches the ground, participants move their hands or dominant limb to maintain balance.
Change in single leg stance time with eye closed | Baseline to end of the 8-week intervention and to end of 8-week follow-up period.
  The maximum amount of time participants are able to maintain stance on their dominant limb with the non-dominant limb flexed 90 degrees and hands held on the waist and with their eyes closed. The test is stopped when the non-dominant limb touches the ground, participants move their hands or dominant limb to maintain balance.
Change in percentage of time spent in sedentary activity. | Baseline to end of the 8-week intervention and to end of 8-week follow-up period.
  Tri-axial accelerometry will be used to determine physical activity over three days (including one weekend day). Child-specific cutoff equations will be used to determine times of sedentary behaviour. Total time in mins will be divided by total wear time to get percentage of time in sedentary activity.
Change in percentage of time spent in moderate to vigorous activity. | Baseline to end of the 8-week intervention and to end of 8-week follow-up period.
  Tri-axial accelerometry will be used to determine physical activity over three days (including one weekend day). Child-specific cutoff equations will be used to determine times spent in moderate to vigorous physical activity. Total time in mins will be divided by total wear time to get the percentage of time in moderate to vigorous activity.
Change in total vector magnitude counts | Baseline to end of the 8-week intervention and to end of 8-week follow-up period.
  Tri-axial accelerometry will be used to determine physical activity over three days (including one weekend day). Vector magnitude counts are a total raw measure of movement.
Change in quality of life score. | Baseline to end of the 8-week intervention and to end of 8-week follow-up period.
  Previously validated Paediatric Quality of Life (PedsQL; physical function section only) will be completed on a 5-point Likert scale and scored. Items are reversed, scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. If more than 50% of the items in the scale are missing, the scale scores should not be computed; mean score = Sum of the items over the number of items answered. A higher score denotes a better quality of life whilst a lower score suggests a poorer quality of life.
Change in pain reported now | Baseline to end of the 8-week intervention and to end of 8-week follow-up period.
  Previously validated paediatric pain questionnaire visual analogue scale for present pain. 10cm (100mm) visual analogue scales from 0 (Not hurting / No discomfort / No pain) to 10 (100) (Hurting a whole lot / Very uncomfortable / Severe pain). The value will be presented as mm from 0. A higher value means greater pain is present.
Change in worst pain | Baseline to end of the 8-week intervention and to end of 8-week follow-up period.
  Previously validated paediatric pain questionnaire visual analogue scale for worst pain in last seven days.10cm (100mm) visual analogue scales from 0 (Not hurting / No discomfort / No pain) to 10 (100) (Hurting a whole lot / Very uncomfortable / Severe pain). The value will be presented as mm from 0. A higher value means greater pain is present.
Change in physical activity enjoyment scale | Baseline to end of the 8-week intervention and to end of 8-week follow-up period.
  Previously validated 16-item 5-point Likert scale from 1 (I disagree a lot) to 5 (I agree a lot). Negatively worded sites are reverse scored, and the overall enjoyment for physical activity score is determined by summing all items. A higher score means greater enjoyment of physical activity.
Change in basic psychological needs in exercise scale score | Baseline to end of the 8-week intervention and to end of 8-week follow-up period.
  Previously validated 18-item 5-point Likert scale from 1 (I disagree a lot) to 5 (I agree a lot). An average score for each subdivision of autonomy, competence, relatedness and teacher relatedness is calculated. A higher score means positive support felt for each subdivision.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Mahaffey, PhD, Principal Investigator — St. Mary's University, Twickenham
Locations (3):
- United Kingdom (3):
  - Orchard Primary school, Hounslow, Greater London
  - Isleworth Town Primary School, Isleworth, Greater London
  - Beavers Primary School, Hounslow, London

IPD SHARING:
Plan to Share IPD: No